CLINICAL TRIAL: NCT01133132
Title: ICCS Directed Physical Activity Enhancement for Colon Cancer Survivors
Brief Title: Interactive Cancer Communication System (ICCS) Directed Physical Activity Enhancement for Colon Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); M.D. Anderson Cancer Center (Other); Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: M-2009-1127; XP08218 (Other: University of Wisconsin Carbone Cancer Center); M-2009-1127 (Other: Institutional Review Board); NCI-2011-00776 (Registry Identifier: NCI Trial ID); A195000 (Other: UW Madison); ENGR/INDUSTRIAL ENGR (Other: UW Madison)
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2018-02

CONDITIONS: Colon Cancer
Keywords: Colon cancer patients who have completed treatment
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): This person will receive usual care and a copy of the National Cancer Institute's Facing Forward booklet and the National Cancer Center Network cancer survivor toolbox.
  Interventions: Behavioral: Survivorship CHESS; Other: Control
- Intervention (Experimental): For those subjects randomized to the Survivorship CHESS condition they will receive a smartphone and access to a web based information system that provides access to clinical information about colon cancer treatment, survivorship, exercise planning and tracking functions to allow these subjects to monitor their self defined exercise goals and objectives.
  Interventions: Behavioral: Survivorship CHESS

INTERVENTIONS:
Behavioral: Survivorship CHESS — Once the consent, baseline survey and one week accelerometer data is received by the UW research team subjects will be randomized to one of the two study conditions. Subjects will be notified of their randomization. Subjects randomized to the Survivorship CHESS condition will be offered training on the smartphone and the CHESS system. The project director (and site research coordinators) will provide training on the smartphone either in person or over the phone. Additionally, an online tutorial will be included in the Survivorship CHESS intervention for subjects to refer to as needed. Participants will then be asked to complete four surveys one baseline and then three follow up surveys.
Other: Control — This person will receive usual care and a copy of the National Cancer Institute's Facing Forward booklet and the National Cancer Center Network cancer survivor toolbox.
  Arms: Control

SUMMARY:
This study will develop and test the benefits of a new ICCS (Interactive Cancer Communication System), a mobile Comprehensive Health Enhancement Support System (Survivorship CHESS) in colon cancer survivors. Survivorship CHESS will provide information, tools, and a support system based on our previous work with FRESH START and CHESS, two highly successful interventions that have promoted lifestyle change among cancer patients and survivors. Survivorship CHESS will be designed to help subjects develop 1) competence in information gathering, decision-making, and behaviors they are trying to change, 2) social support systems to help deal with the cancer experience, and 3) autonomy that comes with regaining a sense of control over their lives; this in turn, will help them adopt or maintain healthy lifestyle behaviors and improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I-III loco-regional colon cancer within the previous 12 months with no evidence of recurrence or new cancers. Participants may be recruited at any time after the initial diagnosis (up to 12 months). Baseline data collection will occur no earlier than 6 weeks after completion of adjuvant treatment
* At least 21 years of age
* Able to speak and read English (educational attainment of at lease 6th grade)
* Engaged in physical activities less than 8 metabolic equivalent tasks (METs) per week
* Not Homeless

Exclusion Criteria:

* Pre-existing medical condition(s) that preclude adherence to an unsupervised exercise program which includes subjects with severe orthopedic conditions or scheduled for a hip or knee replacement within six months; paralysis; end-stage renal disease; dementia; as well as subjects who have unstable angina or who have experienced a heart attack; congestive heart failure or pulmonary conditions that require oxygen or hospitalization within six months; or uncorrected vision or hearing problems or other ergonomic conditions that would preclude the use of the smart phone.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
Change in level of physical activity | 6 M intervention period
  To determine whether stage I-III colon cancer survivors who are randomized to Survivorship CHESS, as compared to those who are assigned to usual care, demonstrate significantly greater increases in levels of physical activity from baseline to completion of the intervention (6 M intervention period).

CONTACTS AND LOCATIONS:
Overall Officials: David H Gustafson, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - Hartford Hospital, Hartford, Connecticut
  - University of North Carolina- Chapel Hill, Chapel Hill, North Carolina
  - M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/